CLINICAL TRIAL: NCT03673189
Title: Sensors for HEalth Recording and Physical Activity Monitoring
Acronym: SHERPAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: LTSI-INSERM U1099 (Unknown); CIC-IT 14-14 (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 35RC17_8836
Record Dates: First submitted 2018-06-12; First posted 2018-09-17 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Physical Activity
Keywords: Sensors; Health Recording
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Prospective, monocentric, with healthy volunteers and patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy volunteers (Experimental): Sensors assigned for 3 weeks
  Interventions: Device: sensors
- Patients with arythmic disease or peripheral vascular disease (Experimental): Sensors assigned for 3 weeks
  Interventions: Device: sensors

INTERVENTIONS:
Device: sensors — Acquisition and transmission of exploitable recordings in the public targeted by the DS, that is to say which allow to draw clinical information in relation to the objectives of the DS (detection of the cardiac rhythm): data without artefact (saturation), in a good signal to noise ratio.

SUMMARY:
The SHERPAM project is part of a scientific and technological context which aim is to record, transmit, analyse the physiological parameters of a patient, as well as to record the feedback to the patient and health professional to suggest the best individualised attitude. The questions of SHERPAM are generic. However, two specific applications will be addressed, in which the partners have already acquired some expertise: the recognition and quantification of physical activity with energy expenditure estimation, and the assessment of walking ability in patients with obliterative vascular disease in the lower limbs. Another application concerns the monitoring of the practice of physical activity and some biological signs in subjects with cardiovascular risk and in cardiac patients (arrhythmogenic diseases). Despite various clinical contexts and health goals, a common approach will be developed.

DETAILED DESCRIPTION:
To assess the SHERPAM Device (DS) by the continuous acquisition and transmission of data (accelerations, rotations, alterations in thoracic volume, heart rate, electrocardiogram) in a real life physical activity practice (subjects in their living environment and during their usual physical practices) using the DS's real-time communication tools, automatic data processing, and the DS's ability to produce information.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers Healthy active subjects aged 50 or over (ie without diagnosed disease, without chronic treatment) and recruited in the sports associations of Ille et Vilaine (cycle tourism clubs).

  * having benefited from an oral or written prescription of physical activity carried out by a health professional and applying this prescription daily in autonomy or in a sports club.

Common to all subjects

* physically active (adherent to a club or sports association or practicing independently according to the recommendations of their physician);
* practicing at least once a week;
* residence located less than 100 km return from Rennes University Hospital
* affiliate or beneficiary of a social protection scheme;
* having given his written consent

Exclusion Criteria:

Common to all subjects

* wearing a pacemaker or implanted cardiac defibrillator (precaution because using telemetry);
* participation in another research protocol;
* persons aver 18 yrs-old subject to legal protection (legal safeguards, guardianship, tutorship), persons deprived of their liberty;
* pregnant or nursing woman.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2019-09-12 (Actual)

PRIMARY OUTCOMES:
asses the continuous acquisition of data by sensors | every day (during 3 weeks)
  transmission and reception of physiological parameters of a patient

SECONDARY OUTCOMES:
Test acceptability of SHERPAM Device | after 7 days of use
  questionnary
Test acceptability of Sherpam Device | after 21 days of use
  questionnary
Test usability of Sherpam Device | after 7 days of use
  questionnary
Test usability of Sherpam Device | after 21 days of use
  questionnary

CONTACTS AND LOCATIONS:
Overall Officials: Carre François, MD, Principal Investigator — Rennes University
Locations (1):
- Unité de Biologie et médecine du Sport, Rennes, Brittany Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Houssein A, Ge D, Gastinger S, Dumond R, Prioux J. Estimation of respiratory variables from thoracoabdominal breathing distance: a review of different techniques and calibration methods. Physiol Meas. 2019 Apr 3;40(3):03TR01. doi: 10.1088/1361-6579/ab0b63. PMID 30818285
- [Result] Dumond R, Gastinger S, Rahman HA, Le Faucheur A, Quinton P, Kang H, Prioux J. Estimation of respiratory volume from thoracoabdominal breathing distances: comparison of two models of machine learning. Eur J Appl Physiol. 2017 Aug;117(8):1533-1555. doi: 10.1007/s00421-017-3630-0. Epub 2017 Jun 13. PMID 28612121
- [Result] Khreis S, Ge D, Rahman HA, Carrault G. Breathing Rate Estimation Using Kalman Smoother With Electrocardiogram and Photoplethysmogram. IEEE Trans Biomed Eng. 2020 Mar;67(3):893-904. doi: 10.1109/TBME.2019.2923448. Epub 2019 Jun 17. PMID 31217092